CLINICAL TRIAL: NCT06625164
Title: The Effects of Core Stabilization Exercises on Respiratory Functions, Trunk Muscle Endurance and Postural Stabilization in Individuals Taking Basic Acting Education,
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Feyza Sule BADILLI HANTAL, Asst.Prof, Yeditepe University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Yeditepe UniversityU
Record Dates: First submitted 2024-04-24; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects
Keywords: core,basic acting education,respiratory functions
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): diaphragm training exercises within the scope of basic acting education;The control group was evaluated at the beginning and at the end of the study.
- exercise group (Active Comparator): diaphragm training exercises within the scope of basic acting education and Planned exercises started to be implemented after one session of training. Exercise group was given exercises by the physiotherapist for 8 weeks, two days a week, during 45 minutes before the acting lessons started.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — core stabilization exercises
  Arms: exercise group

SUMMARY:
The aim of the study is to investigate the effects of a 8-week, core stabilization exercise program on respiratory functions, muscle trunk endurance and postural stabilization in individuals taking basic acting education. The main question it aims to answer is:

the effects of a 8-week, core stabilization exercise program on respiratory functions, muscle trunk endurance and postural stabilization in individuals taking basic acting education

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of a 8-week, core stabilization exercise program on respiratory functions, muscle trunk endurance and postural stabilization in individuals taking basic acting education. The respiratory functions were assessed by the spirometer. Trunk muscle endurance was assessed by Fleksor Trunk Endurance Test (FTET), Biering Sorenson Test (BST) and Lateral Bridge Test (LBT). Postural stabilization was evaluated by Flamingo Balance Test (FBT) and Y Balance Test (YBT). The participants were randomly divided into two groups as Exercise Group (EG) and Control Group (CG) . Both people in EG and CG were taken diaphragmatic training program according to BAE. The core stabilization exercise program was administered for EG, twice a week, 45 minutes a day and for a 8-week duration.

ELIGIBILITY:
The inclusion criterias of this study are;

* Being volunteer
* whose ages between 18-40 years
* whose taking basic acting education course at DC Kozmos Art Academy

Volunteers were excluded from the study if the following conditions will be presented:

* chronic respiratory disease,
* back pain within the last two months,
* pregnancy,
* refusal to sign the informed consent document.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test. Forced vital capacity (FVC) | through study completion, an average of 1 year
  Pulmonary Function Test assessed with spirometer Contec™ SP10W Hand-Held Spirometer according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.It was carried out properly . Forced vital capacity (FVC)
Pulmonary Function Test. Forced expiratory volume at 1st second (FEV1) | through study completion, an average of 1 year
  Pulmonary Function Test assessed with spirometer Contec™ SP10W Hand-Held Spirometer according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.It was carried out properly . Forced expiratory volume at 1st second (FEV1)
Pulmonary Function Test. ratio (FEV1 / FVC) | through study completion, an average of 1 year
  Pulmonary Function Test assessed with spirometer Contec™ SP10W Hand-Held Spirometer according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.It was carried out properly . Tiffeneau ratio (FEV1 / FVC)
Pulmonary Function Test. Peak expiratory flow rate (PEF) | through study completion, an average of 1 year
  Pulmonary Function Test assessed with spirometer Contec™ SP10W Hand-Held Spirometer according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.It was carried out properly . Peak expiratory flow rate (PEF) values
Trunk Muscles Endurance. Trunk Flexors Endurance Test | through study completion, an average of 1 year
Trunk Muscles Endurance. Biering-Sorenson Test | through study completion, an average of 1 year
Trunk Muscles Endurance. Lateral Bridge Test | through study completion, an average of 1 year
Assessment of Postural Stabilization | through study completion, an average of 1 year
  Flamingo balance test

CONTACTS AND LOCATIONS:
Overall Officials: feyza Sule BADILLI HANTAL, PhD, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When the study is registered IPD can be shared with whom contacts with the investigators
Supporting Information: Study Protocol
Time Frame: when trail number is registered and for 5 years
Access Criteria: study protocol will be shared when asked from the investigators